CLINICAL TRIAL: NCT03089164
Title: Assessing the Influence of Postural Changes During Right Heart Catheterization for the Evaluation of Pulmonary Hypertension
Brief Title: Postural Changes During Right Heart Catheterization
Status: Terminated | Type: Observational
Why Stopped: Recruitment challenges and difficulties performing upright hemodynamic measurements using current cath lab setup lead to termination.
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: 16-0554
Record Dates: First submitted 2017-03-20; First posted 2017-03-24 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Pulmonary Hypertension; Right Heart Failure Due to Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Heart Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Right heart catheterization — Each patient will have variables measured supine, sitting and standing positions

SUMMARY:
Hemodynamic measurements obtained during pulmonary artery catheterization are essential for the diagnosis and classification of pulmonary hypertension. Traditionally, right heart catheterization (RHC) is done in the supine position. Cardiac output is known to change significantly based on position, due to the effects of gravity on venous return. There has not been a systematic investigation into these postural effects on pulmonary arterial pressures nor their effect on the diagnosis of pulmonary hypertension. It is our intent to study the differences in measurements obtained during RHC when the patient is supine, seated, and standing.

DETAILED DESCRIPTION:
The investigators also plan a prospective study of patients referred for pulmonary artery catheterization at the UNC cardiac catheterization lab for evaluation of known or suspected pulmonary hypertension. The purpose of this portion of the study is to evaluate the degree to which digital reading of pulmonary artery pressure (PAP) and pulmonary capillary wedge pressure (PCWP) impact the diagnosis and classification of pulmonary hypertension specifically in patients being evaluated for pulmonary hypertension while being tested in the supine, sitting and standing positions.

The investigators will identify 60 patients referred for right heart catheterization to evaluate known or suspected pulmonary hypertension. Patients will have right heart catheterization performed by the clinician that was planning on performing the procedure and a pulmonary hypertension specialist in the Division of Pulmonary and Critical Care Medicine or Division of Cardiology. After informed consent is obtained, the subject will be prepped and draped per protocol in the UNC Cath lab. Their internal jugular vein will be visualized by ultrasound and accessed with a pulmonary artery catheter using standard procedure which also uses fluoroscopy to ensure correct placement of the catheter. Once pressure measurements are obtained from the cardiac chambers and pulmonary arteries, the catheter will be secured into place with tegaderm to allow for mobilization of the patient. The patient will then be asked to sit up on the side of the cath table and the pressure transducer will be re-calibrated to be at the level of the patient's right atrium. Repeat measurements will be obtained of the pulmonary artery and PCWP in this position. After, the patient will be asked to stand up and the pressure transducer once again re-calibrated to estimate the level of the right atrium; new measurements will be obtained in the standing position. Each position will be maintained for 5 minutes before measurements are taken. The supine position measurement will be used for clinical decision making purposes as per usual. The investigators will collect each measurement over at least 10 cardiac cycles and use the mean end-expiratory values to ensure precision.

Once all measurements are obtained, the patient will be asked to return to the supine position. The tegaderm will be released and the catheter removed during sustained expiration maneuver per standard protocol.

No sedation will be administered to the patients.

No further contact will be done with the study subject for the purpose of this research trial.

ELIGIBILITY:
Inclusion Criteria:

* All patients that are 18 years or older regardless of gender or race,
* are referred for RHC for evaluation of possible Pulmonary Arterial Hypertension (PAH)
* provide informed consent

Exclusion Criteria:

* Inability to obtain pulmonary artery pressure or PCWP

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be a cohort of patients referred for right heart catheterization for workup of pulmonary arterial hypertension.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-01-29 (Actual); Study Completion 2018-01-29 (Actual)

PRIMARY OUTCOMES:
Measurement of mean PAP in three positions | During a single right heart catheterization procedure (total time averaging around 30 minutes), about 5 minutes for each position will be needed to obtain each value
  Mean pulmonary arterial pressure pressure (mPAP) will be measured in supine, sitting and standing positions in each subject during a single right heart catheterization procedure
Measurement of PCWP in three positions | During a single right heart catheterization procedure (total time averaging around 30 minutes), about 5 minutes for each position will be needed to obtain each value
  Pulmonary capillary wedge pressure (PCWP) will be measured in supine, sitting and standing positions in each subject during a single right heart catheterization procedure

CONTACTS AND LOCATIONS:
Overall Officials: Hubert "Jimmy" Ford, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No